CLINICAL TRIAL: NCT05484115
Title: Randomized Controlled Clinical Trial on the Application of Heli-FX EndoAnchors in Conjunction With the Endurant II/IIs Endograft in Infrarenal Aortic Aneurysms With a Wide Infrarenal Neck (HERCULES Trial)
Brief Title: Comparison of EVAR and ESAR for Infrarenal Aortic Aneurysms With a Wide Proximal Neck
Acronym: HERCULES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1968
Record Dates: First submitted 2022-07-06; First posted 2022-08-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: AAA; Endovascular treatment; Wide proximal neck; EndoAnchors; Infrarenal; EVAR (Endovascular aneurysm repair); ESAR (Endosuture aneurysm repair); Endurant II/IIs stent graft system; Heli-FX EndoAnchor system
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Intervention Model Description: HERCULES is a post-market, prospective, global, multicenter, randomized (1:1), two-arm, superiority trial designed to compare ESAR to standard EVAR clinical outcomes in treatment of infrarenal AAA in patients having wide proximal aortic neck diameters (≥ 28mm and ≤ 32mm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard endovascular aneurysm repair (EVAR) using the Endurant II/IIs stent graft system (Active Comparator)
  Interventions: Device: endovascular aneurysm repair (EVAR) using the Endurant II/IIs stent graft system
- Endosuture aneurysm repair (ESAR) with the Endurant II/IIs in conjunction with Endoanchors (Active Comparator)
  Interventions: Device: endosuture aneurysm repair (ESAR) using Heli-FX EndoAnchor system

INTERVENTIONS:
Device: endovascular aneurysm repair (EVAR) using the Endurant II/IIs stent graft system — treatment of AAA's with wide proximal neck diameters with Endurant II/IIs endograft system
  Arms: Standard endovascular aneurysm repair (EVAR) using the Endurant II/IIs stent graft system
Device: endosuture aneurysm repair (ESAR) using Heli-FX EndoAnchor system — treatment of AAA's with wide proximal neck diameters with the Endurant II/IIs in conjunction with the Heli-FX EndoAnchor system
  Arms: Endosuture aneurysm repair (ESAR) with the Endurant II/IIs in conjunction with Endoanchors

SUMMARY:
The HERCULES trial is a Randomized controlled clinical trial designed to prospectively compare endosuture aneurysm repair (ESAR) to standard endovascular aneurysm repair (EVAR) clinical outcomes in treatment of infrarenal abdominal aortic aneurysm (AAA) in subjects having wide proximal aortic neck diameters (≥ 28mm and ≤ 32mm).

DETAILED DESCRIPTION:
HERCULES is an investigator driven trial and a collaborative research project with Medtronic.

Design; Prospective, post-market, global, multicenter, randomized (1:1), two-arm, superiority trial

Up to 300 subjects will be recruited in up to 40 sites in Europe and the US. All subjects shall be followed per local societal guidelines and per the Endurant II/IIs and Heli-FX EndoAnchor instruction for use (IFU) recommendations for post-implant follow-up and CT-imaging, with expected assessments at baseline, index procedure(s), 1-month, and annually at 1, 2, 3, 4, and 5 years post-index procedure.

Devices used in HERCULES include the Endurant II/IIs stent graft system (EVAR arm) and the Endurant II/IIs stent graft system plus the Heli-FX EndoAnchor System (ESAR arm)

This study is being conducted to collect clinical evidence from treatment of patients with infrarenal AAA having wide proximal aortic neck diameters (≥ 28mm and ≤ 32mm), comparing clinical outcomes with treatment of the AAA with the Endurant II/IIs stent graft in conjunction with Heli-FX EndoAnchors to treatment of the AAA with the Endurant II/IIs stent graft alone. Though both the Endurant II/IIs stent graft and Heli-FX EndoAnchors are commercially approved in this indication, clinical evidence comparing these two treatments in patients with wide proximal aortic neck diameters is not currently available. Collecting clinical data specific to this patient population, including procedure and imaging data as well as long term outcomes, will provide a foundation to further characterize the clinical outcomes of treatment for patients with infrarenal AAA with wide proximal aortic neck diameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Provided written informed consent
* Clinical necessity for treatment of the AAA, according to the current guidelines in the geographies participating
* Elective repair
* Eligible anatomy for treatment with the Endurant II/IIs stent graft system and Heli-FX EndoAnchor system according to the IFU of both devices
* Infrarenal neck diameter ≥ 28 mm and ≤32 mm
* Proximal neck length ≥10mm

Exclusion Criteria:

* Anatomy outside the IFU of the ndurant II/IIs stent graft system and Heli-FX EndoAnchor system
* Planned use of AUI main body device
* Patient is participating in another clinical study, potentially conflicting with the outcomes of the current study.
* Patient with eGFR < 30 ml/min/1.73m2 before the intervention
* Patient's life expectancy <2 years as judged by the investigator
* Patient has a psychiatric or other condition that may interfere with the study
* Patient has a known allergy to any device component
* Patients with a systemic infection who may be at increased risk of endovascular graft infection.
* Patient has a coagulopathy or uncontrolled bleeding disorder
* Patient has a ruptured, leaking, or mycotic aneurysm
* Patient is not eligible for standard EVAR
* Patient had a Cerebro Vascular Accident (CVA) or a myocardial infarction (MI) within the prior three months
* Patient is pregnant (Female patients of childbearing potential only)
* Patient has active COVID-19 infection or has been diagnosed with long COVID-19 requiring hospitalization within the 6 months prior to procedure.
* Patient has previously been treated with stent grafts in the aorto-iliac arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2033-04 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint at on proximal seal outcomes | 1 year follow-up
  The primary endpoint is a composite endpoint based on core lab reported data from computed tomography (CT) with contrast imaging of freedom from:
  1. type IA endoleak and
  2. Migration of the proximal portion of the stent graft ≥5 mm (compared to 1-month imaging) and
  3. Aneurysm sac growth ≥5 mm (compared to 1-month imaging).

SECONDARY OUTCOMES:
Freedom from type IA endoleak | 1 year follow-up
  Freedom from type IA endoleak
Freedom from migration | 1 year follow-up
  Migration of the proximal portion of the stent graft ≥5 mm (compared to 1-month imaging)
Freedom from aneurysm sac growth | 1 year follow-up
  Aneurysm sac growth ≥5 mm (compared to 1-month imaging).
Freedom from neck dilatation ≥ 3 mm | 1 year follow-up
  Neck dilatation ≥ 3 mm (compared to 1-month imaging).

CONTACTS AND LOCATIONS:
Overall Officials: MMPJ Reijnen, Prof. Dr., Principal Investigator — Rijnstate, Arnhem, the Netherlands; K. Donas, Prof. Dr., Principal Investigator — Asklepios Clinic Langen, Langen, Germany
Locations (36):
- United States (15):
  - Washington Regional Medical Center, Washington, Arkansas
  - Mt Sinai Med Ctr, Miami Beach, Florida
  - Loyola, Maywood, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Beaumont University Hospital, Royal Oak, Michigan
  - Alina Health, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Robert Wood Johnson University Medical Center, New Brunswick, New Jersey
  - Sisters of Charity hospital, Buffalo, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - NC Heart& Vascular, Raleigh, North Carolina
  - Promedica Toledo Hospital, Toledo, Ohio
  - Ballad Health/Holston Valley, Kingsport, Tennessee
  - Virginia Commonwealth University (VCU), Richmond, Virginia
- France (3):
  - HCL Lyon, Lyon
  - Saint Joseph Marseille, Marseille
  - Les Franciscaines, Nîmes
- Germany (3):
  - Asklepios Klinik Langen, Langen, Hesse
  - Universitatsklinikum Frankfurt, Frankfurt
  - University Hospital Leipzig, Leipzig
- Italy (2):
  - IRCCS Ospedale Policlinico San Martino, Genova, Metropolitan City of Genoa
  - Osp. S.Orsola Malpighi - Bologna, Bologna
- Netherlands (4):
  - Noordwest ziekenhuis, Alkmaar, North Holland
  - Spaarne Gasthuis, Haarlem, North Holland
  - Rijnstate hospital, Arnhem
  - Catharina Ziekenhuis, Eindhoven
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Ramon Y Cajal, Madrid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- EHC-Hôpital de Morges, Morges, Switzerland
- United Kingdom (4):
  - Queen Elizabeth University Hospital, Glasgow, Glasgow
  - Leeds General Infirmary, Leeds
  - St. George's Hospital, London
  - St. Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: No